CLINICAL TRIAL: NCT05676645
Title: Pharmacokinetics of Drugs Used to Treat Uncomplicated Malaria in Breastfeeding Mother-infant Pairs: An Observational Pharmacokinetic Study
Brief Title: Pharmacokinetics of Antimalarials in Breastfeeding Ugandan Mother-infant Pairs
Acronym: MILK Malaria
Status: Active, not recruiting | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Makerere University (Other); Malawi-Liverpool-Wellcome Clinical Research Programme (Unknown)
Responsible Party: Principal Investigator, Catriona Waitt, Professor Catriona Waitt, University of Liverpool
Other Study IDs: MILK Malaria
Record Dates: First submitted 2022-12-13; First posted 2023-01-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples will be stored for up to 5 years for analysis of additional measures related to the protocol objectives
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Breastfeeding women who have been prescribed (by a clinician independent from the study team) artemether-lumefantrine to treat uncomplicated malaria
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Artemether-lumefantrine — National policy recommendation for treatment of uncomplicated malaria in Uganda

SUMMARY:
Lactating women requiring treatment for uncomplicated malaria will be identified and invited for sampling. The decision to treat them with first-line treatment will have been made by the clinician, not by a member of the study team. The study team will not make any adjustments to the prescribed treatment. Artemether-lumefantrine comprises six doses of medication, with the initial two doses given 8 hours apart on Day 1, and dosing 12-hourly on Day 2 and Day 3. Intensive pharmacokinetic sampling will be undertaken after Dose 5, as indicated in the schema under Section 5: plasma and breastmilk samples will be obtained pre-dose and at 2, 4, 6, 8 hours after dose. In addition, sparse sampling will be undertaken on either of these occasions; at pre-dose and between 1 to 6 hours after the first dose; a trough (pre-dose) sample after the Dose 3 or Dose 4 and lastly at 5, 7, and up to 14-days after the first dose. A heelprick sample will also be obtained from the breastfed infants at maternal trough (prior to maternal dose) and at a random timepoint (once per infant) over the 8-hour pharmacokinetic sampling visit to characterize concentrations of these drugs over an 8-hour dosing interval. In addition, a single heelprick sample will be obtained from the infant whenever the mother returns after treatment for the late sampling time points (5, 7, and 14 days post the first dose). Due to the long half-life of lumefantrine of approximately 6 days plasma sampling will be performed up to day 14 to characterise the terminal elimination of the drug. Concentrations of total plasma and breastmilk lumefantrine and desbutyl-lumefantrine will be determined.

DETAILED DESCRIPTION:
The endpoints of this study relate to the amount of antimalarial drug present in maternal blood, breastmilk and infant blood. The study is not powered for antimalarial efficacy, and therefore formal assessment of parasitological clearance is not required. The participants will be followed up until 30-40 days after completion of antimalarial therapy, and if recurrent symptoms occur, management will be as clinically indicated. Details regarding further clinical investigations and management required by either mother or infant during the follow-up period will be recorded on the CRF.

ELIGIBILITY:
Inclusion Criteria:

1. A personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
2. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Woman is aged 18 years or older, and mothers between the age of 14-17, who are considered emancipated minors.
4. Receiving treatment for uncomplicated malaria
5. Breastfeeding at enrolment

Exclusion Criteria:

1. Severe maternal or infant illness which in the opinion of the patient's clinician would interfere with her participation in the study
2. Breastfed infant is aged over 12 months
3. Partner objection to participate in the study
4. Maternal objection to infant participation

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ugandan breastfeeding women requiring treatment for uncomplicated malaria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
AUC0-24 of lumefantrine in maternal plasma and breastmilk | 0-24 hours after dose
  Maternal plasma exposure of lumefantrine
AUC0-24 of lumefantrine breastmilk | 0-24 hours after dose
  Breastmilk exposure of lumefantrine
Milk to plasma ratio of lumefantrine | 0-24 hours after dose
  Ratio of AUC in breastmilk to maternal plasma

SECONDARY OUTCOMES:
AUC desbutyl-lumefantrine plasma | 0-24 hours after dose
  Plasma exposure of active metabolite
AUC desbutyl-lumefantrine breastmilk | 0-24 hours after dose
  Breastmilk exposure of active metabolite
Milk to plasma ratio of desbutyl-lumefantrine | 0-24 hours after dose
  Ratio of breastmilk to maternal plasma of active metabolite
Infant concentration lumefantrine | 0-8 hours after maternal dose
  Infant lumefantrine exposure
Infant concentration desbutyl-lumefantrine | 0-8 hours after maternal dose
  Infant exposure to active metabolite
Infant development | 0-1 year old
  Infant assessment using Gross Motor Development Score (IGMDS)
Depression and anxiety in mothers | 0-1 year postpartum
  Patient Health Questionnaire (PHQ9)
Depression and anxiety in mothers | 0-1 year postpartum
  General Anxiety Disorder (GAD7)
Maternal beliefs about medicines | 0-1 year postpartum
  Beliefs about Medicines questionnaire (BMQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data showing age, number of weeks postpartum and drug concentrations in plasma, breastmilk and infant plasma will be made available for future use following primary publication.
Supporting Information: Study Protocol
Time Frame: After primary publication - intention is to place anonymised data on drug concentrations on an online repository such as Zenodo
Access Criteria: Weblink not yet available.